CLINICAL TRIAL: NCT04577690
Title: Pectoral Nerve (PECS) Block for Cardiac Implantable Electronic Devices (CIED) Implantation Surgery
Brief Title: PECS Study for CIED Implantation Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Katherine Taylor, Associate Professor, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000065122
Record Dates: First submitted 2020-09-28; First posted 2020-10-08 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Pain, Postoperative; Child; Adolescent
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Intervention Model Description: Using a computer-generated table, patients will be randomized to one of two groups: PECS block or Local infiltration only. Group allocation are concealed in sealed, opaque, sequentially numbered envelopes that are opened on the day of surgery.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The nursing staff in the post anesthesia care unit, patient and outcome assessors will be blinded to the patient allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PECS block (Experimental): A PECS block of 0.25 % bupivacaine with epinephrine 1:200000 (below the toxic dose limit of 3 mg/kg) in divided doses to cover the fascial planes identified in PECS I and PECS II. At the completion of surgery, the wound will be infiltrated with up to 0.2 ml/kg of 0.25 % bupivacaine into the wound.
  Interventions: Drug: Bupivacaine 0.25% with epinephrine 1:200000 by PECS block and wound infiltration
- Infiltration (Active Comparator): At the completion of surgery, the EP cardiologist will infiltrate the wound with up to 0.8 ml/kg of 0.25 % bupivacaine with epinephrine 1:200000.
  Interventions: Drug: Bupivacaine 0.25% with epinephrine 1:200000 by wound infiltration only

INTERVENTIONS:
Drug: Bupivacaine 0.25% with epinephrine 1:200000 by PECS block and wound infiltration — The anesthesiologist will administer bupivacaine 0.25% with epinephrine 1:200000 by PECS block after induction of anesthesia before surgical incision. The EP cardiologist will also administer bupivacaine 0.25% with epinephrine 1:200000 by infiltrating the wound after surgery is complete.
  Other Names: PECS block
  Arms: PECS block
Drug: Bupivacaine 0.25% with epinephrine 1:200000 by wound infiltration only — The EP cardiologist will administer Bupivacaine 0.25% with epinephrine 1:200000 by infiltrating the wound after surgery is complete.
  Other Names: Infiltration
  Arms: Infiltration

SUMMARY:
We aim to determine whether pectoral nerve block (PECS) performed after induction of anesthesia but before surgical incision results less opioid use in the post operative period compared with local infiltration alone in children undergoing Cardiac Implantable Electronic Device (CIED) surgery.

DETAILED DESCRIPTION:
The current anaesthetic management of CIED surgery at Sickkids is local anaesthetic infiltration by the EP cardiologist or a Pectoral nerve block (PECS) on an ad-hoc basis depending on the anaesthesiologist on a case by case basis. It is not known whether one technique provides better post- operative pain control and fewer adverse events than the other. In either case, the patient receives opioids as required during and after the procedure. Patients typically go home with a prescription for opioids to be taken for the first few days after surgery.

The PECS block is a recognized effective anaesthetic technique used for both intraoperative and postoperative pain control in adult breast surgery, chest wall procedures as well as one case report for CIED implantation and a small series in paediatric cardiac surgery. The advantages of the PECS block in these surgical procedures includes improved analgesia and reduced opioid use.

The investigators plan to conduct an RCT with two groups.

Group 1 will receive a PECS block (using 0.8 ml/kg of 0.25% bupivacaine with epinephrine 1: 200000 divided in two equal volumes between the two planes) by the anaesthesiologist and local infiltration (up to 0.2 ml/kg of 0.25% bupivacaine with epinephrine 1:200000) by the surgeon.

Group 2 will receive local infiltration (up to 0.8 ml/kg 0.25 % bupivacaine with epinephrine 1:200000) by the surgeon alone.

Both groups will be given opioids as rescue analgesics as deemed necessary during their procedure and as rescue analgesia postoperatively, so that no patient will have untreated pain.

ELIGIBILITY:
Inclusion Criteria:

• All patients 3-18 years undergoing CIED surgery in the chest

Exclusion Criteria:

* Children < 3 years of age at time of procedure as bupivacaine is not licensed for this age group.
* No parental or patient consent
* Allergy to bupivacaine
* Pregnancy or lactation
* Any condition or diagnosis, that could in the opinion of the Principal Investigator or delegate interfere with the participant's ability to comply with study instructions, might confound the interpretation of the study results, or put the participant at risk.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative morphine consumption | 0 hours
  Amount of morphine or morphine equivalents used after surgery

SECONDARY OUTCOMES:
Severity of pain | 0 hours, 6 hours, 12 hours and at discharge from hospital
  Severity of pain will be measured using and Numerical Rating Score (NRS) or Face, Legs, Activity, Cry and Consolability (FLACC) score as appropriate for age.
Incidence of nausea/emesis postoperatively | Until discharge from recovery room, assessed up to 2 days
  Any self-reported episodes of nausea and any emesis will be recorded
Incidence of pruritus | Until discharge from recovery room, assessed up to 2 days
  Any self-reported episodes of pruritus will be recorded.
Adverse events | Until discharge from recovery room, assessed up to 2 days
  Any occurrence of hematoma, pneumothorax, lung injury or local anesthesia toxicity will be recorded
Time to discharge from recovery room | Until discharge from recovery room, assessed up to 2 days
  Time from admission to recovery room to discharge from recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Taylor, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Froyshteter AB, Bhalla T, Tobias JD, Cambier GS, Mckee CT. Pectoralis blocks for insertion of an implantable cardioverter defibrillator in two patients with Duchenne muscular dystrophy. Saudi J Anaesth. 2018 Apr-Jun;12(2):324-327. doi: 10.4103/sja.SJA_624_17. PMID 29628849
- [Background] Fujiwara A, Komasawa N, Minami T. Pectoral nerves (PECS) and intercostal nerve block for cardiac resynchronization therapy device implantation. Springerplus. 2014 Aug 5;3:409. doi: 10.1186/2193-1801-3-409. eCollection 2014. PMID 25120950
- [Background] Al Ja'bari A, Robertson M, El-Boghdadly K, Albrecht E. A randomised controlled trial of the pectoral nerves-2 (PECS-2) block for radical mastectomy. Anaesthesia. 2019 Oct;74(10):1277-1281. doi: 10.1111/anae.14769. Epub 2019 Jul 4. PMID 31273773
- [Background] Altiparmak B, Korkmaz Toker M, Uysal AI, Turan M, Gumus Demirbilek S. Comparison of the effects of modified pectoral nerve block and erector spinae plane block on postoperative opioid consumption and pain scores of patients after radical mastectomy surgery: A prospective, randomized, controlled trial. J Clin Anesth. 2019 May;54:61-65. doi: 10.1016/j.jclinane.2018.10.040. Epub 2018 Nov 3. PMID 30396100
- [Background] Amir A, Jolin S, Amberg S, Nordstrom S. Implementation of Pecs I and Pecs II Blocks as Part of Opioid-Sparing Approach to Breast Surgery. Reg Anesth Pain Med. 2016 Jul-Aug;41(4):544-5. doi: 10.1097/AAP.0000000000000401. No abstract available. PMID 27315180
- [Background] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971
- [Background] Blanco R. The 'pecs block': a novel technique for providing analgesia after breast surgery. Anaesthesia. 2011 Sep;66(9):847-8. doi: 10.1111/j.1365-2044.2011.06838.x. No abstract available. PMID 21831090
- [Background] Kumar KN, Kalyane RN, Singh NG, Nagaraja PS, Krishna M, Babu B, Varadaraju R, Sathish N, Manjunatha N. Efficacy of bilateral pectoralis nerve block for ultrafast tracking and postoperative pain management in cardiac surgery. Ann Card Anaesth. 2018 Jul-Sep;21(3):333-338. doi: 10.4103/aca.ACA_15_18. PMID 30052231